CLINICAL TRIAL: NCT06908044
Title: Effectiveness of Bryophyllum Pinnatum in the Treatment of Primary Dysmenorrhea: a Prospective Observational Study
Brief Title: Assessing the Therapeutic Potential of a Traditional Botanical Remedy for Menstrual Pain: Insights From a Prospective Observational Analysis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK-2024-01549
Record Dates: First submitted 2025-04-01; First posted 2025-04-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Dysmenorrhea Primary
Keywords: Bryophyllum Pinnatum; Primary Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group with Bryophyllum Pinnatum (Experimental): The study group receive Bryophyllum Pinnatum (tablets) for 6 Months
  Interventions: Drug: Bryophyllum

INTERVENTIONS:
Drug: Bryophyllum — Bryophyllum Pinnatum - tablets, for 6 Months

SUMMARY:
Primary dysmenorrhea (PDM) affects round 60 to 90% of women and has a great impact on everyday life of affected women, leading to decreased work productivity, cognitive activity and cuts in social life. The aetiology of pain symptoms mainly results from increased contractile activity. Non-rhythmic and uncoordinated contractions lead to high uterine pressure, which together with vasoconstriction result in reduced blood flow and ultimately in painful uterine ischemia. Conventional treatment options are limited to pain medication such as paracetamol, non-steroidal anti-inflammatory drugs (NSAID) or - especially, but not only, if contraception is also desired - hormonal contraceptives. Due to the frequent occurrence of (sometimes severe) side effects, there has been a lack of effective treatment options that can be taken regularly without hesitation. The succulent herb Bryophyllum pinnatum (BP) (Lam.) Oken. (Crassulaceae) (synonym: Kalanchoe pinnata) originated in Madagascar,but is at present found in wide-ranging (sub)tropical regions of Africa and Asia. In Switzerland, BP is often used in obstetrics and gynaecology, so far mainly for preterm labour (as a tocolytic), and in some cases for overactive bladder syndrome, nocturia and sleeping disorders, but not for dysmenorrhea. Current pharmacological data on the inhibition of myometrial contractile mechanisms by BP preparations as well as its reported use against inflammation and pain in ethnomedicine made us hypothesize that BP might be a new treatment option for PDM.

Primary objective of the study:

Assessment of the PDM - associated menstrual pain

Secondary objectives of the study:

Assessment of the quality of life in PDM Recording of AEs under study medication Compliance

ELIGIBILITY:
Inclusion Criteria

* Age between 18 and 45 years with regular menstrual cycles (21-35 days)
* Menstrual pain rated 6 or higher on an 11-point PI-NRS during the most painful day
* In good general health
* Provided written informed consent
* Willing to maintain the same personal hygienic product throughout the study (e.g., tampons, pads, menstrual cups; no changes in menstrual hygiene practices allowed during the study)

Exclusion Criteria

* Secondary dysmenorrhea (i.e. in endometriosis, adenomyosis, urogenital malformations)
* Currently taking, or had taken in the past two months, hormonal forms of birth control
* Dysmenorrhea reasonably suspected to be due to a IUD
* Prior or current liver or kidney disease, inflammatory bowel disease, reproductive cancer (uterine, ovarian, etc.)
* Personal history of known hypersensitivity to the used drug or its ingredients or to drugs with a similar chemical structure
* Other diseases that do not allow the subject to assess the nature and scope as well as possible consequences of the clinical study
* Pregnant or breastfeeding women
* Signs that the subject is unlikely to comply with the protocol (e.g., unwillingness to cooperate)
* Alcohol/drug abuse
* Non-German speaking patients (Patient information is only available in German)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Score (Numeric Rating Intensity - NRI) | From enrollment to the end of treatment at 6 months
  Measurement of the intensity of the pain during the menstrual periods: a score of 0 means no pain, a score of 10 means the maximal pain

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Private Centre for Obstetrics and Gynecology "Geburt und Familie", Aarau, Canton of Aargau
  - Paracelsus Zentrum am Grossmünster, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the primary and secondary outcomes of each patients undergone treatment with Bryophyllum Pinnatum
Supporting Information: ICF
Time Frame: from the end of the study (31/12/2028) for 10 years
Access Criteria: Researchers who want to reaserch further Bryophyllum Pinnatum in Dysmenorrhea or related research topics. They can contact the PI to receive information. They will receive the row data of the outcomes of each patient.

REFERENCES:
- [Background] Zurfluh L, Spinelli MG, Betschart C, Simoes-Wust AP. Repurposing of Bryophyllum pinnatum for dysmenorrhea treatment: a systematic scoping review and case series. Front Pharmacol. 2023 Dec 1;14:1292919. doi: 10.3389/fphar.2023.1292919. eCollection 2023. PMID 38130407